CLINICAL TRIAL: NCT03014050
Title: Effectiveness of Bio-Electro Stimulation Therapy for the Treatment of Motor and Non-Motor Symptoms in Parkinson's Disease - A Pilot Study
Brief Title: Bio Electro Stimulation Therapy for Parkinson's Disease
Acronym: BEST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Karin Schon, Assistant Professor, Anatomy & Neurobiology, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-34609; BEST-PD2017 (Other: Boston Medical Center)
Record Dates: First submitted 2016-12-12; First posted 2017-01-09 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Parkinson Disease
Keywords: physical activity; fitness; cognition; mood; depression; anxiety; sleep quality; tremor; gait
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Tremor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EH: Stimulation of Head Point (Experimental): Electrical stimulation of the head point of the hand (EH, experimental stimulation); intervention with e-Tapper TT-R1
  Interventions: Device: e-Tapper TT-R1
- CS: Control Stimulation (Active Comparator): Electrical stimulation of the leg point of the hand (CS, control stimulation); intervention with e-Tapper TT-R1
  Interventions: Device: e-Tapper TT-R1

INTERVENTIONS:
Device: e-Tapper TT-R1 — The e-Tapper is a non-invasive, handheld electronic device designed to apply micro current stimulation to a person's hands at specified points representing various body parts, such as the head, leg, or foot. This is one form of "Bio-Electro Stimulation Therapy" known as the "11-point Hand Treatment System". The current delivered is less than one milliampere.

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor dysfunction and non-motor symptoms. Here, the investigators propose in a pilot device feasibility trial to examine whether "Bio Electro Stimulation Therapy" (B.E.S.T.) with a small, non-invasive, handheld electronic device designed to apply micro current stimulation to a person's hand can ameliorate some of the symptoms of PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor dysfunction, cognitive impairment, and other non-motor symptoms. Here, we propose to use "Bio Electro Stimulation Therapy" (B.E.S.T.) using the "e-Tapper TT-R1"owned by Immumax International Co. Ltd., a Hong Kong based company. The "e-Tapper" is a non-invasive, handheld electronic device designed to apply micro current stimulation to a person's hand at specified points representing various body parts, such as the head, leg, or foot. This is one form of Bio Electro Stimulation Therapy, known as "11-point Hand Treatment System". The current delivered is less than one milliampere. Anecdotal evidence suggests that this micro current stimulation may reduce resting tremor, restore facial expressions, and improve ease of movement, mood, and sleep quality in patients with PD. Scientific evidence for the effectiveness of the B.E.S.T. Hand Therapy appears to be lacking in the English language (Western) literature. The goal of this pilot device feasibility study is to examine whether B.E.S.T. can increase physical activity and functional fitness, enhance cognition, improve mood and subjective sleep quality, and modulate resting tremor and gait parameters in PD patients over a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* High functioning without presence of cognitive impairment or dementia
* Native-English speaker or fluent in English
* Diagnosis of Parkinson's disease (Hoehn & Yahr stages I-III)

Exclusion Criteria:

* Implanted medical devices, such as a pacemaker or defibrillator
* Prescription medication or other drugs that affect the brain (e.g. anti-depressants, anxiolytics), except prescription medication for the treatment of Parkinson's disease
* Poor vision that cannot be corrected with glasses or contact lenses
* Presence of musculoskeletal impairments (e.g. fractures, hemiplegia, chronic joint pain)
* Not being able to walk without assistance
* Diagnosis of dementia or mild cognitive impairment
* Diabetes mellitus
* Taking medications for diabetes mellitus
* Skin irritation, disease or wound on the hands
* Current heart conditions, such as congestive heart failure, tachycardia, or other arrhythmias
* History of heart attack
* Psychiatric or neurological disorders other than Parkinson's disease (e.g. Major Depressive Disorder, anxiety disorder, epilepsy)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Physical activity | 10-12 weeks
  Assessment of physical activity with body-worn sensor
Visuospatial Cognition | 10-12 weeks
  Assessment of visuospatial cognition
Mood | 10-12 weeks
  Mood will be assessed with questionnaires.
Sleep quality | 10-12 weeks
  Sleep quality will be assessed with a questionnaire.
Resting tremor | 10-12 weeks
  Resting tremor will be assessed with body-worn sensors.
Gait | 10-12 weeks
  Gait will be assessed with body-worn sensors.

SECONDARY OUTCOMES:
Perceived pain | 10-12 weeks
  Perceived pain will be assessed with a questionnaire.
Quality of life and subjective health status | 10-12 weeks
  This questionnaire, called "The 39-Item Parkinson's Disease Questionnaire" (PDQ-39) assesses how often people with Parkinson's disease experience difficulties in their lives in several domains, including mobility, activities of daily living, emotional well-being, stigma, social support, perceived cognition, communication, and bodily discomfort. A "PDQ-39 Summary Index" score will be calculated. Scores range from 0 (best quality of life) to 100 (worst quality of life).
Physical activity - Other | 10-12 weeks
  Subjective physical activity will be assessed with a questionnaire.
Functional Fitness | 10-12 weeks
  Participants will undergo short field tests of functional fitness.
Cognition - Language | 10-12 weeks
  Assessment of verbal fluency
Cognition - Cognitive Control | 10-12 weeks
  Assessment of executive functions
Cognition - learning and memory | 10-12 weeks
  Assessment of learning and memory

CONTACTS AND LOCATIONS:
Overall Officials: Karin Schon, Ph.D., Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No